CLINICAL TRIAL: NCT02558179
Title: Prospective Multicenter Cross Sectional Study of the American International Biotechnology (AIBiotech) Gynecologene Test for the Evaluation of Bacterial Vaginosis/Vaginitis in Symptomatic Women
Brief Title: Diagnosing Bacterial Vaginosis/Vaginitis (BV) Using the Gynecologene Test Method
Acronym: SAGE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: American International Biotechnology (Industry)
Responsible Party: Sponsor
Other Study IDs: SAGE-001
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Vaginosis, Bacterial
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples With DNA — Extracted DNA from vaginal swab(s) will be maintained after evaluation for a time period up to 1 year.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Nugent Score >/= 7: Signs and symptoms of vaginitis/vaginosis, including vaginal discharge, pruritis, irritation, and/or dyspareunia. Diagnosis of bacterial vaginosis (study group) according to Nugent score and/or diagnosis of vulvovaginal candidiasis; and/or diagnosis of Trichomonas vaginalis.
- Nugent Score< 7: Signs and symptoms of vaginitis/vaginosis, including vaginal discharge, pruritis, irritation, and/or dyspareunia. Bacterial vaginosis not diagnosed according to Nugent score (<7).

SUMMARY:
This study is designed as a prospective evaluation of the diagnostic performance of the multiplex nucleic acid-based genetic test (Gynecologene Next-Generation Sequencing test) to identify known significant causative organisms in bacterial vaginosis/vaginitis and other major pathogens and normal commensals in symptomatic women during the reproductive years. Vaginal fluid samples will be split and tested with the comparator methods and Nugent score, with the results evaluated according to sensitivity, specificity, positive predictive value, and negative predictive value. Laboratorians performing each test will be blinded to the clinical history and any prior test results to minimize ascertainment bias.

Each subject will be followed routinely for up to 6 weeks after initial visit for vaginosis/vaginitis by telephone or office visit at the discretion of the treating physician.

DETAILED DESCRIPTION:
Bacterial vaginosis (BV, or vaginal bacteriosis) and vaginitis are the most common vaginal infections of women during the child-bearing years, with BV alone accounting for 27-41% 1 prevalence in Americans. BV is characterized by replacement of the healthy lactobacillus-dominant microbiome by a diverse polymicrobial overgrowth of multiple taxa of commensal facultative anaerobes and other pathogenic bacteria. Molecular-based phylogenetic analyses, including the newly-completed Human Microbiome Project and other next-generations sequencing (NGS) studies, revealed the complexity of the vaginal microbiome in health and disease. BV does not appear to be a single entity, but rather consists of multiple bacterial community clusters. Clusters are dominated by Lactobacillus iners, Lactobacillus crispatus, or anaerobic combinations with or without Lactobacillus spp. (species) in varying proportions. In addition, multiple significant BV-associated pathogens were discovered that had escaped notice with other detection methods such as cultures; previously overlooked were Atopobium vaginae, Lactobacillus iners and other Lactobacillus spp., and multiple Lachnospiraceae spp (Bacterial Vaginosis Associated 1, Bacterial Vaginosis Associated 2, and Bacterial Vaginosis Associated 3; BVA1, BVA2 and BVA 3 respectively). This multisite study proposes to evaluate the sensitivity and specificity of the Gynecologene Next-Generation Sequencing test in women with symptoms of vaginitis/vaginosis. To the investigators' knowledge, the Gynecologene is the first commercially-available comprehensive NGS-based laboratory-developed test available to assist with diagnosis and clinical management of BV.

This multisite site study compares the diagnostic performance of the Gynecologene Next-Generation Sequencing test with the clinical diagnosis of bacterial vaginosis/vaginitis (Nugent score). The second objective is to compare the sensitivity and specificity of the Gynecologene Score with the Nugent Score for diagnosis of bacterial vaginosis/vaginitis. The third objective is to identify the prevalence and diagnostic thresholds of bacterial loads with the Gynecologene test.

Women between 18-55 years of age will be eligible for this study when diagnosed with bacterial vaginosis or vaginitis confirmed using the CDC (Centers for Disease Control) diagnostic gold standard of Nugent score; Amsel criteria will also be recorded. Other inclusion as well as exclusion criteria exist. A minimum of 5 geographically different sites will be enrolled in the study. Co-investigators will follow the protocol to enroll participants and collect 2 vaginal swabs and 1 slide smear. The patient has no financial gain nor responsibility within this protocol.

Overall, the study will have 90% power at a significance level of 0.05 to detect ± 5% positive percent agreement of the study device with the predicate device. To achieve this level of power, 100 total samples will be assayed per group to account for withdrawals and treatment failures. Samples that contain more than one targeted organism can be counted twice as the analyses for each organism are independent of each other. The provision of treatment, including type, dose, and duration, is solely at the discretion of the clinician according to his/her current routine procedures to reflect typical contemporary practice.

AIBiotech will serve as a central medical diagnostic laboratory for this trial. Results of all analytical tests will be provided to the Principal Investigator.

Data for analysis will be blinded for patient identification and other PHI (protected health information) by the study administrator. Data will be analyzed and reported.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age and any race (African-American, Hispanic, Asian/Pacific Islander, native American, white).
* Women during reproductive years prior to menopause and in no case over age 55 years.
* Signed Informed Consent document obtained prior to the initiation of screening procedures.
* Signs and symptoms of vaginitis/vaginosis, including vaginal discharge, pruritis, irritation, and/or dyspareunia.
* Diagnosis of bacterial vaginosis (study group) according to Nugent score (see below); and/or diagnosis of vulvovaginal candidiasis; and/or diagnosis of Trichomonas vaginalis.
* Clinical Diagnosis: Nugent Score: The presence of abnormal vaginal flora at initial diagnosis confirmed by gram stain, with all subjects with BV (bacterial vaginosis or bacterial vaginitis) having Nugent score > 7.
* Inclusion Criteria of Control Group: same as Study Group, but Nugent Score < 7.
* No active major medical or psychological problems that could be complicated by study participation.

Exclusion Criteria:

* Treatment with any investigational prescription product within 28 days of study screening.
* Post-menopausal or greater than 55 years of age.
* Prior history of hysterectomy or vaginal surgery.
* Prior or currently active autoimmune disease requiring management with systemic immunosuppression for any reason. Such conditions include inflammatory bowel disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-related thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatological disease.
* Any infection requiring parenteral/ enteral antibiotic therapy or causing fever (body temperature > 100.5°F or 38.1°C) within 4 weeks prior to study screening.
* Any medical intervention or other condition which, in the opinion of the Physician-Investigator could compromise adherence with study requirements or otherwise compromise study subject safety and the study's objectives.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women at least 18 years of age will be eligible for this study when diagnosed with bacterial vaginosis or vaginitis confirmed using the CDC (Centers for Disease Control) diagnostic gold standard of Nugent score; Amsel criteria will also be recorded.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Evidence of Confirmed BV Through Next Generation Sequencing Gynecologene Assay | 2 weeks after receiving sample
  Vaginal swabs meeting inclusion criteria will be assessed for BV using the Gynecologene Assay. Confirmation of BV.

SECONDARY OUTCOMES:
Comparison of Sensitivity of Gynecologene to Clinical Diagnosis of BV by Nugent Score (Gold Standard) | 2 weeks after receving sample
  calculation of Sensitivity of the condition of BV (true positive rate) using Gynecologene assay as the "test" and Nugent Score as the "gold standard"
Comparison of Specificity of Gynecologene to Clinical Diagnosis of BV by Nugent Score (Gold Standard) | 2 weeks after receving sample
  calculation of Specificity of the condition of BV (true negative rate) using Gynecologene assay as the "test" and Nugent Score as the "gold standard"

OTHER OUTCOMES:
Bacterial Load | 3 months
  identify the prevalence and diagnostic thresholds of bacterial loads found with each specimen using the Gynecologene test. All bacteria will be included and will use the vaginal microbiome to assign specific bacteria. Load will be reported as a percentage of individual bacteria to the total amount found in that sample. Since all samples are unbiquie - identifying every bacteria is not possible. All organisms that have reached the threshold coverage limit within the assay will be reported. Threshold limits are defined within the validation of the Gynecologene assay

CONTACTS AND LOCATIONS:
Overall Officials: David G Bostwick, MD, Study Director — American International Biotechnology (AI Biotech)
Locations (4):
- United States (4):
  - David Greenspan OB-GYN, Phoenix, Arizona
  - Desert Jewel Obstetrics and Gynecology, Scottsdale, Arizona
  - Daniel McDyer OB-GYN, Jacksonville, Florida
  - Unified Clinical Research, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Klebanoff MA, Turner AN. Bacterial vaginosis and season, a proxy for vitamin D status. Sex Transm Dis. 2014 May;41(5):295-9. doi: 10.1097/OLQ.0000000000000124. PMID 24722382
- [Background] Taylor BD, Darville T, Haggerty CL. Does bacterial vaginosis cause pelvic inflammatory disease? Sex Transm Dis. 2013 Feb;40(2):117-22. doi: 10.1097/OLQ.0b013e31827c5a5b. PMID 23324974
- [Background] Mitchell C, Manhart LE, Thomas K, Fiedler T, Fredricks DN, Marrazzo J. Behavioral predictors of colonization with Lactobacillus crispatus or Lactobacillus jensenii after treatment for bacterial vaginosis: a cohort study. Infect Dis Obstet Gynecol. 2012;2012:706540. doi: 10.1155/2012/706540. Epub 2012 May 30. PMID 22693410
- [Background] Swidsinski A, Loening-Baucke V, Swidsinski S, Verstraelen H. Polymicrobial Gardnerella biofilm resists repeated intravaginal antiseptic treatment in a subset of women with bacterial vaginosis: a preliminary report. Arch Gynecol Obstet. 2015 Mar;291(3):605-9. doi: 10.1007/s00404-014-3484-1. Epub 2014 Sep 23. PMID 25245669
- [Background] Parma M, Stella Vanni V, Bertini M, Candiani M. Probiotics in the prevention of recurrences of bacterial vaginosis. Altern Ther Health Med. 2014 Winter;20 Suppl 1:52-7. PMID 24473986
- [Background] Marrazzo JM, Thomas KK, Fiedler TL, Ringwood K, Fredricks DN. Relationship of specific vaginal bacteria and bacterial vaginosis treatment failure in women who have sex with women. Ann Intern Med. 2008 Jul 1;149(1):20-8. doi: 10.7326/0003-4819-149-1-200807010-00006. PMID 18591634
- [Background] Marrazzo JM. Interpreting the epidemiology and natural history of bacterial vaginosis: are we still confused? Anaerobe. 2011 Aug;17(4):186-90. doi: 10.1016/j.anaerobe.2011.03.016. Epub 2011 Apr 16. PMID 21524714
- [Background] Muzny CA, Sunesara IR, Griswold ME, Kumar R, Lefkowitz EJ, Mena LA, Schwebke JR, Martin DH, Swiatlo E. Association between BVAB1 and high Nugent scores among women with bacterial vaginosis. Diagn Microbiol Infect Dis. 2014 Dec;80(4):321-3. doi: 10.1016/j.diagmicrobio.2014.09.008. Epub 2014 Sep 16. PMID 25262105
- [Background] Wang B, Xiao BB, Shang CG, Wang K, Na RS, Nu XX, Liao Q. Molecular analysis of the relationship between specific vaginal bacteria and bacterial vaginosis metronidazole therapy failure. Eur J Clin Microbiol Infect Dis. 2014 Oct;33(10):1749-56. doi: 10.1007/s10096-014-2128-5. Epub 2014 May 10. PMID 24816815
- [Background] Aagaard K, Petrosino J, Keitel W, Watson M, Katancik J, Garcia N, Patel S, Cutting M, Madden T, Hamilton H, Harris E, Gevers D, Simone G, McInnes P, Versalovic J. The Human Microbiome Project strategy for comprehensive sampling of the human microbiome and why it matters. FASEB J. 2013 Mar;27(3):1012-22. doi: 10.1096/fj.12-220806. Epub 2012 Nov 19. PMID 23165986
- [Background] Srinivasan S, Hoffman NG, Morgan MT, Matsen FA, Fiedler TL, Hall RW, Ross FJ, McCoy CO, Bumgarner R, Marrazzo JM, Fredricks DN. Bacterial communities in women with bacterial vaginosis: high resolution phylogenetic analyses reveal relationships of microbiota to clinical criteria. PLoS One. 2012;7(6):e37818. doi: 10.1371/journal.pone.0037818. Epub 2012 Jun 18. PMID 22719852
- [Background] van de Wijgert JH, Borgdorff H, Verhelst R, Crucitti T, Francis S, Verstraelen H, Jespers V. The vaginal microbiota: what have we learned after a decade of molecular characterization? PLoS One. 2014 Aug 22;9(8):e105998. doi: 10.1371/journal.pone.0105998. eCollection 2014. PMID 25148517